CLINICAL TRIAL: NCT06656390
Title: A First-in-Human, Open-Label, Multi-Center Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ALK201 for Injection in Adult Participants With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Antitumor Activity of ALK201 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Allink Biotherapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALK201-01
Record Dates: First submitted 2024-10-20; First posted 2024-10-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Advanced Cancer; Advanced Solid Tumors
Keywords: First-in-human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A: Dose-escalation Phase, Part B: Dose-expansion Phase (Experimental): A dose-escalation study to determine the MTD and the subsequent doses for dose expansion study (Part B).
  A dose-expansion study which will enroll the select indications.
  Interventions: Drug: ALK201

INTERVENTIONS:
Drug: ALK201 — Administered intravenously, once every 3 weeks

SUMMARY:
This is a first-in-human (FIH), open-label, multicenter dose escalation and expansion study of ALK201. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of ALK201 as a monotherapy in adult participants with Advanced Solid Tumors. The study will also identify recommended dose(s) for subsequent clinical studies of ALK201.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 and ≤75 years old on the day of signing the ICF
* At least 1 measurable lesion per RECIST v1.1
* Expected survival ≥3 months
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1
* Adequate organ function
* Female participants of childbearing potential or male participants whose partner is a female of childbearing potential agree to use medically effective contraceptive methods from the date of signing the ICF until at least 6 months after the last dose of the IP, and during this period, male participants are not allowed to donate sperms

Exclusion Criteria:

* Active or pre-existing autoimmune diseases that may relapse
* Pleural effusion, pericardial effusion, or intraperitoneal effusion accompanied with clinical symptoms, clinically poorly controlled, or requiring repeated drainage
* Allergies to any component of ALK201 or other monoclonal antibodies
* Primary central nervous system malignancies, or active metastases to central nervous system and/or metastases to meninges
* Combined with ≥ Grade 2 stomatitis and/or nose bleeding at screening
* Vaccinated with live vaccines within 4 weeks prior to the first dose

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-10-22 (Estimated); Study Completion 2028-04-22 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ALK201 in adult participants with advanced solid tumors; To determine the maximum tolerated dose (MTD); To determine the recommended dose(s) of ALK201 for subsequent clinical studies. | Approximately 36 months
  Dose-limiting toxicity (DLT); The incidence and severity of treatment-emergent adverse events (TEAEs) and treatment-related adverse events (TRAEs) according to CTCAE v5.0.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of ALK201. | Approximately 36 months
  PK parameters after single and multiple doses: area under the concentration-time curve from time zero to the last measurement (AUC0-last)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: area under the concentration-time curve from time zero to infinity (AUC0-inf)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: Maximum serum Concentration (Cmax)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: Time to Maximum Concentration(Tmax)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: trough Concentration(Ctrough)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: Clearance(CL)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: apparent Distribution Volume(Vd)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: steady-state apparent distribution volume (Vss)
To evaluate the pharmacokinetics (PK) of ALK201 | Approximately 36 months
  PK parameters after single and multiple doses: terminal half-life (t1/2)
To evaluate the immunogenicity of ALK201. | Approximately 36 months
  The generation of anti-drug antibodies (ADAs).
To evaluate the preliminary antitumor activity of ALK201 | Approximately 36 months
  Objective Response Rate (ORR)
To evaluate the preliminary antitumor activity of ALK201 | Approximately 36 months
  Duration of Response (DOR)
To evaluate the preliminary antitumor activity of ALK201 | Approximately 36 months
  Disease Control Rate (DCR)
To evaluate the preliminary antitumor activity of ALK201 | Approximately 36 months
  Progression-Free Survival (PFS)
To evaluate the preliminary antitumor activity of ALK201 | Approximately 36 months
  Overall Survival (OS)
To evaluate the biomarkers. | Approximately 36 months
  Descriptive analysis will be made to describe the correlation between clinical outcomes and FGFR2 genetic alterations.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Care Wollongong, Wollongong, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided